CLINICAL TRIAL: NCT03474276
Title: A Multi-center, Randomized Controlled Comparison of Three Renutrition Strategies for the Management of Moderate Acute Malnutrition Among Children From 6 to 24 Months (Madagascar, Niger, Central African Republic and Senegal)
Brief Title: Comparing Several Strategies to Manage Moderate Acute Malnutrition Among Children From 6 to 24 Months Old
Acronym: MALINEA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Collaborators: Action Contre la Faim (Other); Centre de Recherches Médicales et Sanitaires CERMES Niger (Unknown); Institut Pasteur de Madagascar (Other); Institut Pasteur de Bangui (Ambiguous); Institut Pasteur de Dakar (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-062; FPC N° 2013-4025 (Other Grant/Funding Number: Ministère de l'Europe et des Affaires Etrangères)
Record Dates: First submitted 2016-06-13; First posted 2018-03-22 (Actual); Last update posted 2022-05-24 (Actual); Status verified 2022-05

CONDITIONS: Moderate Acute Malnutrition
Keywords: Children; Africa; Metagenomic; Prebiotic; Randomized Controlled Trial; Pragmatic trial; Azithromycin; Cognitive impairment
MeSH Terms: conditions — Cognitive Dysfunction | interventions — Azithromycin; Anti-Bacterial Agents; fructooligosaccharide; Prebiotics; Albendazole; Antiparasitic Agents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): Fortified Blended Flour (in association with a single dose of Albendazole at inclusion for children older than 12 months).
  200 grams / day for children between 6 and 11 months. 300 grams / day for children aged from 12 to 24 months old.
  Interventions: Drug: Albendazole; Dietary Supplement: Fortified blend flour
- Azythromycin (Active Comparator): Fortified Blended Flour (in association with a single dose of Albendazole at inclusion for children older than 12 months) associated to Azythromycin, 20mg/kgs/days during the three first days of the study.
  Interventions: Drug: Azythromycin; Drug: Albendazole; Dietary Supplement: Fortified blend flour
- Prebiotic (Active Comparator): Fortified Blended Flour mixed with Inuline and fructo-oligosaccharides (Synergy1) 2g/day, given to the child through the whole intervention (in association with a single dose of Albendazole at inclusion for children older than 12 months)
  Interventions: Dietary Supplement: Inuline and fructo-oligosaccharides; Drug: Albendazole; Dietary Supplement: Fortified blend flour

INTERVENTIONS:
Drug: Azythromycin — Administration of azythromycin to the child at inclusion (3 days) 20 mgs/kgs/day : three days
  Other Names: Antibiotics
  Arms: Azythromycin
Dietary Supplement: Inuline and fructo-oligosaccharides — Administration of inuline and fructo-oligosaccharides (Synergy1) 2g/day, mixed with the fortified blend flour given to the child through the whole intervention.
  Other Names: Prebiotic
  Arms: Prebiotic
Drug: Albendazole — Administration of Albendazole at inclusion of the child : 200mgs, one administration
  Other Names: Antiparasitic drug
Dietary Supplement: Fortified blend flour — Children from 6 to 11 months : 200 grams / day Children from 12 to 24 months : 300 grams / day
  Compostion of the fortified blend flour per 100 grams : either :
  Mil (whole grains): 58,56 g/100g, Soybeans (fat meal): 16,54g/100g Peanuts (roasted seeds): 8,75g/100g, Cane sugar: 7,35 g/100g Whole milk (Powder): 7,56g/100g, MSV MAM: 0,28g/100g, iodized salt :0,45g/100g, CaC03: 0,48g/100g,Amylase BAN: 0,03g/100g OR Corn (whole grains): 53,29g/100g, Soybeans (dry seeds): 17,82g/100g, Peanuts (roasted seeds): 9,00 g/100g, Cane sugar: 11,00 Whole milk (Powder): 5,00g/100g, Soybean Oil (Purified): 1,24g/100g, Peanut oil (Purified): 1,13g/100g, MSV MAM: 0,27g/100g, iodized salt: 0,53 g/100g, Ca3(PO4)2: 0,62g/100g, KCl: 0,09g/100g
  Other Names: Lacteal flour

SUMMARY:
The aim of this open-label randomized controlled trial conducted in four African countries (Madagascar, Niger, Central African Republic and Senegal) is to compare three strategies of renutrition for moderate acute malnutrition (MAM) in children based on modulation of the gut microbiota with enriched flours alone, enriched flours with prebiotics or enriched flours coupled with antibiotic treatment. Cognitive development of children (Senegal) will also be studied and compared.

DETAILED DESCRIPTION:
The main objective of this study is to improve the nutrition strategy used to take in charge moderate acute malnutrition (MAM) which is the major milestone before severe malnutrition. This will be based on the modulation of the gut microbiota with adjunct product added to standard nutrition flours.

The purpose of the MALINEA study is to compare three management strategies for Moderate Acute Malnutrition (MAM) in children aged between 6 months and 2 years old on recovery defined by a weight/size gain at 3 months.

The 3 groups will be compared on several anthropometric measurements [Weight, length, Mid Upper Arm Circumference (MUAC)], clinical characteristics, adherence and tolerance to interventions between before and after a 3 months intervention Cognitive development of children (Senegal) will also be studied and compared, at inclusion, 3 months and 6 months after inclusion.

The investigators will also investigate the microbiomes of malnourished children at inclusion and at 3 and 6 months after inclusion to compare it to the ones of normonourished children.

ELIGIBILITY:
Inclusion Criteria:

* Children aged from 6 to 24 months olds.
* Moderate acute malnutrition defined by a -3 ≤ Weight/Height z-score < -2 SD.
* Written informed consent of parents or legal guardian.
* Child able to be brought back to the centre on the two following days of inclusion.
* Child able to be followed up during at least three months.

Exclusion Criteria:

* Severe malnutrition defined by a mid upper arm circumference < 115 mm OR Weight/Height z-score < -3 SD OR presence of nutritional oedema.
* Clinical complications or according to the physician any clinical sign requiring care outside of the recruitment centre (referral to specialised centre or hospitalisation)
* Diarrhea with mucus and bloody stools.
* Current incompatible treatment : Antacids, Cetirizine, Digoxin, Ergotamine, Azidothymidine.
* Known hypersensitivity to macrolides or albendazole (or one of its components)
* Known allergy to enriched flours or prebiotics used in the study, or one of its components.

Ages: 6 Months to 24 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1357 (Actual)
Dates: Start 2018-01-31 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
Recovery at three month | Three month
  Recovery at three months, defined by: Weight/Size Z-score ≥ -1.5 SD measured at 2 following consultations without hospitalization, transfer, death or lost to follow up

SECONDARY OUTCOMES:
Cognitive-motor development (Senegal) | Baseline, three, six and nine months after inclusion
  Developmental Milestones Checklist II (DMC II) questionnaire to evaluate participating children cognitive and motor abilities.
Comparison of the Operational Taxonomic Unit composition of stool samples according to the nutritional status | Baseline, three and six months after inclusion
  Each sample will be ADN extracted using Quiagen technology 16S and 18S amplification will be conducted following Hughert et al. (2014) and Tang et al. (2015). PCR products will be sequenced using NGS Illumina plateform. Sequences will be analyzed using Mothur 1.37.6 software and Silva data base (https://www.arb-silva.de/browser). OTU (Operational Taxonomic Unit) composition will be determined for each sample.
  OTU composition of samples from well and malnourished children will be compared using mann whitney test, and shift in OTUs during renutrition will be analysed using survival analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Ronan JAMBOU, PhD, Principal Investigator — Institut Pasteur; Muriel Vray, phD, Principal Investigator — Institut Pasteur
Locations (4):
- Institut Pasteur de bangui - Centre Nutritionnel de Gbangouma et Centre de Santé Saint-Joseph, Bangui, Central African Republic
- Institut Pasteur de Madagascar - CRENAM Andohotapenaka et Centre de Santé Mitia, Antananarivo, Madagascar
- Centre de santé intégré ACF de Tchake et d'Issawanne, Maradi, Niger
- Institut Pasteur de Dakar - Poste de Santé Hamo V, Dakar, Guédiawaye, Senegal

REFERENCES:
- [Derived] Vray M, Hedible BG, Adam P, Tondeur L, Manirazika A, Randremanana R, Mainassara H, Briend A, Artaud C, von Platen C, Altmann M, Jambou R. A multicenter, randomized controlled comparison of three renutrition strategies for the management of moderate acute malnutrition among children aged from 6 to 24 months (the MALINEA project). Trials. 2018 Dec 4;19(1):666. doi: 10.1186/s13063-018-3027-3. PMID 30514364
- See also: GRET: French development NGO fighting poverty and inequalities, providing solutions for development [150 projects per year in 30 countries] — http://www.gret.org/
- See also: Institut Pasteur: Private non-profit foundation whose mission is to prevent and treat diseases through research, teaching, and public health initiatives. — http://www.pasteur.fr/en
- See also: Action contre la faim [Action against hunger] : International humanitarian organization providing communities with access to safe water and sustainable solutions to hunger. — http://www.actionagainsthunger.org